CLINICAL TRIAL: NCT02460380
Title: The Effects of Vitamin D Supplementation on Transforming Growth Factor-beta1 and Vascular Endothelial Growth Factor in Vitamin D-Deficient Women With Polycystic Ovary Syndrome: A Randomized Placebo-Controlled Trial
Brief Title: The Effects of Vitamin D on Angiogenic Factors in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Richard Grazi, Director of Genesis Fertility and Reproductive Medicine, Obstetrics and Gynecology, Maimonides Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-06-03
Record Dates: First submitted 2015-05-23; First posted 2015-06-02 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: Polycystic Ovary Syndrome; Vitamin D Deficiency
MeSH Terms: conditions — Polycystic Ovary Syndrome; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 (Active Comparator): Women allocated to vitamin D3 group received one capsule 50.000 IU of vitamin D3 once weekly for eight weeks.
  Interventions: Drug: Vitamin D3
- Placebo (Placebo Comparator): Women in the placebo group received once capsule of placebo once weekly for eight weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — Women allocated to vitamin D arm received one capsule 50.000 IU of vitamin D3 once weekly for eight weeks.
  Arms: Vitamin D3
Other: Placebo — Women in the placebo arm received once capsule of placebo once weekly for eight weeks
  Arms: Placebo

SUMMARY:
Polycystic Ovary Syndrome (PCOS) affects 5 to 10% of women of reproductive age. It is characterized by a cluster of hyperandrogenism, hyperinsulinemia, menstrual dysfunction, hirsutism and infertility. Although the pathogenesis of PCOS is unknown, accumulating evidence suggests that the dysregulation of some angiogenic factors, such as transforming growth factor-β (TGF-β) and vascular endothelial growth factor (VEGF), may be implicated. TGF-βs and VEGF exert a diverse range of biological functions regulating cell proliferation, angiogenesis, fibroblast activation and tissue fibrosis. PCOS ovaries show all the hallmarks of TGF-β and VEGF upregulation, including increased collagen deposition in ovarian stroma and theca, supported by increased vascularity. Consistent with this, The investigators recently showed that TGF-β1 is increased in serum of PCOS women while its circulating receptor soluble endoglin (sENG) is decreased, resulting in greater TGF-β1 bioavailability. Furthermore, it has been shown that women with PCOS have increased VEGF levels in the serum and/or follicular fluid. PCOS patients also have decreased vitamin D levels, and vitamin D treatment has been previously shown to improve various clinical parameters in PCOS women, including glucose intolerance, hypertension and androgen levels. Interestingly, vitamin D has been shown to decrease TGF-β1 and VEGF levels in several diseases, including myelofibrosis and various human cancer cells. Therefore, the investigators hypothesize that vitamin D treatment of PCOS women will result in a decrease of serum TGF-β1 levels and/or VEGF levels concomitant with improvement in clinical disease parameters. In addition, the investigators hypothesize that improvement in clinical disease parameters will correlate with changes in serum VEGF levels and TGF-β1 bioavailability. Our aim in the present study is to investigate the effects of vitamin D treatment on serum VEGF and TGF-β1/sENG levels in PCOS women, and assess whether changes in these angiogenic factors following vitamin D treatment correlate with clinical disease in these women. For this end, PCOS patients who are vitamin D-deficient will be treated with vitamin D and their serum levels of VEGF, TGF-β1 and its sENG receptor will be measured before and after treatment. In addition, clinical disease parameters will be recorded before and 4 months after treatment, including serum glucose and insulin levels, serum androgen levels, and blood pressure.

The proposed study aims to identify a putative link between vitamin D, VEGF, and TGF-β1 in the context of PCOS, and provide a novel molecular explanation for the beneficial clinical effects of vitamin D on PCOS patients.

DETAILED DESCRIPTION:
This study is a randomized, single blind, placebo-controlled trial to evaluate the effect of vitamin D on vitamin D-deficient women with PCOS. 93 reproductive-aged women diagnosed with PCOS presenting to Maimonides Medical Center for annual check-up between October 2013 and March 2015 were screened for vitamin D deficiency (defined as 25 hydroxy-vitaminD [25OH-D] levels <20 ng/mL). All participants signed the informed consent and the study was approved by the international review board (IRB) of Maimonides Medical Center. PCOS was diagnosed according to the Rotterdam Consensus (ESHRE/ASRM criteria), i.e. the presence of two of three criteria: oligo- or anovulation, signs of clinical hyperandrogenism, and/or biochemical signs of hyperandrogenism and polycystic ovaries on ultrasonography after exclusion of specific identifiable disorders (thyroid disorder, hyperprolactinemia, congenital adrenal hyperplasia, androgen-secreting tumors, and Cushing's syndrome). The investigators included women aged between 18 and 38 years who were not: 1) pregnant, postpartum, breastfeeding, or 2) taking any vitamin D supplements, metformin or any hormonal therapy.

Interventions and blood collection:

68 women diagnosed with PCOS and vitamin D deficiency were enrolled. Participants were allocated to each group according to a computer-generated list using ratio 2/1 (Vitamin D/placebo). Women allocated to vitamin D group received one capsule 50.000 IU of vitamin D3 once weekly for eight weeks. The vitamin D supplementation regimen was extracted from the Endocrine Society guidelines. Women in the placebo group received once capsule of placebo once weekly for eight weeks. The placebo was prepared at Maimonides Medical Center's pharmacy. To ensure compliance, The investigators called each participant once weekly and reminded her to take her pill. Fasting blood samples were collected by venipuncture before starting and within two weeks after completing the treatment (vitamin D or placebo). Blood samples were allowed to clot for 30 minutes at room temperature before centrifugation at 1,200 rpm for 10 minutes. Serum was stored at -80°C in aliquots until assayed.

The assays of all measured hormones, 25OH-D, VEGF, TGF-β1, sENG, and AMH:

Serum 25OH-D levels were measured before and after completing the treatment. The levels were determined by the ADVIA Centaur vitamin D assay (Siemens Healthcare Diagnostics). Dehydroepiandrosterone sulfate (DHEAS), testosterone, sex hormone-binding globulin (SHBG), thyroid-stimulating hormone (TSH), follicle-stimulating hormone (FSH), and luteinizing hormone (LH) were measured using IMMULITE 2000 XPi immunoassay system (Siemens Healthcare USA). Insulin and prolactin concentrations were quantified by DXL 800 immunoassay analyzer according to manufacturer's protocols (Beckman Coulter). Insulin resistance was calculated according to the homeostatic model assessment (HOMA) (29) by using the following formula: Insulin resistance (HOMA IR) = [fasting insulin (µU/mL) x fasting glucose (mmol/L)]/22.5. 17OH-progesterone level was determined by ELISA assay (Eagle BioSciences). AMH concentration was measured using the ultrasensitive AMH/MIS CLIA kit (AnshLabs). TGF-β1 concentration was measured using Human TGF-beta1 Quantikine ELISA kit according to manufacturer's protocols (R&D Systems). sENG levels were quantified by Human Endoglin/CD105 Quantikine ELISA kit (R&D Systems). VEGF concentration was quantified using Human VEGF Quantikine ELISA kit according to manufacturer's protocols (R&D Systems). The inter-assay and intra-assay coefficients of variation for all assays were less than 10%.

Clinical parameters:

All the clinical parameters were evaluated before and four months after the completion of treatment. These parameters included blood pressure (BP), Ferriman-Gallwey score (FGS) (hirsutism score), acne status, and interval between periods.

Statistical analysis:

Data were tested for normality. All values were expressed as mean ± standard error of the mean (SEM). A paired student's t-test was used to compare pre- and post-treatment serum levels and clinical parameters. Correlation between changes in angiogenic factors and changes in clinical disease parameters was analyzed using Pearson's test and linear regression. X2-test was used to evaluate the changes in acne after treatment. SigmaStat (SPSS Science, Chicago, IL) was used for statistical analysis. P<0.05 was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Women with PCOS who have vitamin D deficiency (serum 25-hydroxyvitamin D<20 ng/mL)

Exclusion Criteria:

* Pregnant, postpartum, breast feeding
* Taking Metformin, vitamin D, or any hormonal therapy

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

REFERENCES:
- [Derived] Irani M, Seifer DB, Grazi RV, Julka N, Bhatt D, Kalgi B, Irani S, Tal O, Lambert-Messerlian G, Tal R. Vitamin D Supplementation Decreases TGF-beta1 Bioavailability in PCOS: A Randomized Placebo-Controlled Trial. J Clin Endocrinol Metab. 2015 Nov;100(11):4307-14. doi: 10.1210/jc.2015-2580. Epub 2015 Oct 20. PMID 26485217

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 93 women were screened for vitamin D deficiency. Sixty-eight women were diagnosed with vitamin D deficiency and were included in the study and randomly allocated into the two groups.
Period: Overall Study
Arm/Group | Vitamin D3 | Placebo
Started | 45 | 23
Completed | 35 | 18
Not Completed | 10 | 5
Not completed — Withdrawal by Subject | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D3 | Placebo | Total
Number analyzed (Participants) | 45 | 23 | 68
Age, Continuous [Mean (Standard Deviation); unit: years]
  number analyzed (Participants) | 35 | 18 | 53
  (all) | 30.5 (6.4) | 29.6 (7.6) | 30.2 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  number analyzed (Participants) | 35 | 18 | 53
  Female | 35 | 18 | 53
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 17 | 48
  Not Hispanic or Latino | 14 | 6 | 20
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States: number analyzed (Participants) | 35 | 18 | 53
  United States | 35 | 18 | 53

OUTCOME MEASURES:

1. Primary Outcome: Effect of Vitamin D on Angiogenic Factors
Description: Serum TGF-β1/sENG ratio as a measure of TGF-β1 bioavailability
Time Frame: Baseline (pre-treatment) and 8 weeks later (post-treatment)
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 35 | 18
ratio
  Serum TGF-β1/sENG before treatment | 6.7 (0.4) | 5.6 (0.5)
  Serum TGF-β1/sENG after treatment | 5.9 (0.4) | 5.5 (0.4)

2. Primary Outcome: Effect of Vitamin D on Angiogenic Factors
Description: Serum VEGF level
Time Frame: Baseline (pre-treatment) and 8 weeks later (post-treatment)
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 35 | 18
pg/mL
  Serum VEGF level before treatment | 1106.4 (36.5) | 893.1 (90.2)
  Serum VEGF level after treatment | 965.3 (42.7) | 866 (70.8)

3. Secondary Outcome: The Effects of Vitamin D3 on Clinical Disease Parameters in Women With PCOS
Description: Interval between periods as a measure ovulatory dysfunction
Time Frame: Baseline (pre-treatment) and 4 months later (two months after the completion of treatment)
Measure: Mean (Standard Error); unit: Days
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 35 | 18
Days
  Interval between periods before treatment | 80.2 (9.8) | 79 (9)
  Interval between periods after treatment | 60 (6.7) | 75 (9)

4. Secondary Outcome: The Effects of Vitamin D3 on Clinical Disease Parameters in Women With PCOS
Description: Blood pressure
Time Frame: Baseline (pre-treatment) and 4 months later (two months after the completion of treatment)
Measure: Mean (Standard Error); unit: mmHG
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 35 | 18
mmHG
  Systolic blood pressure before treatment | 112 (1.9) | 113 (2.8)
  Systolic blood pressure after treatment | 108 (1) | 109 (2.3)
  Diastolic blood pressure before treatment | 68.4 (1.1) | 69 (1.7)
  Diastolic blood pressure after treatment | 67.9 (1.3) | 67 (1.6)
  Mean arterial pressure before treatment | 83 (1.2) | 84 (1.9)
  Mean arterial pressure after treatment | 81 (1.1) | 81 (1.7)

5. Secondary Outcome: The Effects of Vitamin D3 on Clinical Disease Parameters in Women With PCOS
Description: The homeostatic model assessment (HOMA) is a method used to quantify insulin resistance. Insulin resistance is a condition in which cells fail to respond to the normal actions of the hormone insulin. The HOMA index was calculated as the product of fasting plasma blood glucose and insulin divided by 22.5.
Time Frame: Baseline (pre-treatment) and 8 weeks later (post-treatment)
Measure: Mean (Standard Error); unit: HOMA IR score
Groups:
- Vitamin D3 Group Before Treatment: Women allocated to vitamin D3 group received one capsule 50.000 IU of vitamin D3 once weekly for eight weeks.
  Vitamin D3: Women allocated to vitamin D arm received one capsule 50.000 IU of vitamin D3 once weekly for eight weeks.
Arm/Group | Vitamin D3 Group Before Treatment | Placebo
Number analyzed (Participants) | 35 | 18
HOMA IR score
  Insulin resistance (HOMA-IR)before treatment | 2.07 (0.37) | 1.58 (0.3)
  Insulin resistance (HOMA-IR) after treatment | 2.03 (0.22) | 1.52 (0.24)

6. Secondary Outcome: The Effects of Vitamin D3 on Clinical Disease Parameters in Women With PCOS
Description: Free testosterone
Time Frame: Baseline (pre-treatment) and 8 weeks later (post-treatment)
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 35 | 18
ng/dL
  Free testosterone before treatment | 0.59 (0.06) | 0.61 (0.08)
  Free testosterone after treatment | 0.68 (0.06) | 0.68 (0.11)

7. Secondary Outcome: The Effects of Vitamin D3 on Clinical Disease Parameters in Women With PCOS
Description: Lipid profile
Time Frame: Baseline (pre-treatment) and 8 weeks later (post-treatment)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 35 | 18
mg/dL
  HDL before treatment | 46 (2.4) | 47 (2.9)
  HDL after treatment | 48 (2.6) | 50 (3.2)
  LDH before treatment | 106 (6.1) | 103 (7.7)
  LDL after treatment | 100 (4.1) | 101 (5.1)
  Total cholesterol before treatment | 183 (6.5) | 179 (9)
  Total cholesterol after treatment | 166 (11) | 177 (6.3)
  Triglycerides before treatment | 138 (22) | 113 (21)
  Triglycerides after treatment | 117 (20) | 98 (13)

8. Secondary Outcome: The Effects of Vitamin D3 on Clinical Disease Parameters in Women With PCOS
Description: Ferriman-Gallwey score is a method used to assess and quantify hirsutism in women. A total score < 8 is considered normal whereas a score of 8 to 15 indicates mild hirsutism. A score >15 indicates moderate or severe hirsutism.
Time Frame: Baseline (pre-treatment) and 4 months later (two months after the completion of treatment)
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 35 | 18
Scores on a scale
  Ferriman-Gallwey score before treatment | 9.8 (1.5) | 8.1 (1.4)
  Ferriman-Gallwey score after treatment | 8.1 (1.5) | 7.6 (1.5)

ADVERSE EVENTS:
Arm/Group | Vitamin D3 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/18
Other Adverse Events (participants affected / at risk) | 0/35 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No